CLINICAL TRIAL: NCT00086138
Title: Depression in Alzheimer's Disease (DIADS-2)
Brief Title: Depression in Alzheimer's Disease-2
Acronym: DIADS-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Constantine G. Lyketsos, Chairman, Bayview Psychiatry, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01MH066136 (NIH); U01MH066136 (NIH); DATR A4-GPX
Record Dates: First submitted 2004-06-25; First posted 2004-06-28 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease; Depression
Keywords: Alzheimer's disease; Depression
MeSH Terms: conditions — Alzheimer Disease; Depression | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive sertraline at a target dose of 100mg daily.
  Interventions: Drug: Sertraline (Zoloft)
- 2 (Placebo Comparator): Participants will receive placebo matched to sertraline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline (Zoloft) — Sertraline: range of 25 to 125 mg per day for 24 weeks
  Arms: 1
Drug: Placebo — Placebo designed to mimic sertraline taken daily for 24 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to learn whether treating individuals with Alzheimer's disease and depression with the anti-depressant medication sertraline (Zoloft) is helpful to people with Alzheimer's disease and to their families and caregivers.

DETAILED DESCRIPTION:
Participants are randomly assigned to treatment with sertraline (range 25-125 mg per day) or identical placebo for 24 weeks. There are 8 scheduled in-person visits in the 24 weeks. Visits include neuropsychological testing. Caregivers are asked to are the patient on a Daily Affect Diary for 6 weeks during the study period. Telephone followup is done at weeks 36 and 48. Both groups receive caregiver support/education.

ELIGIBILITY:
Inclusion:

* Ability of the participant, caregiver or surrogate to provide written informed consent.
* Dementia due to Alzheimer's disease
* Stable treatment for Alzheimer's disease
* Ability for the participant's caregiver to accompany the participant to study visits and participate in the study.

Exclusion

* Presence of a brain disease that might otherwise explain the presence of dementia
* Clinically significant hallucinations or delusions
* Current treatment of antipsychotics, anticonvulsants, and other antidepressants, benzodiazepines, or other psychotropic medications
* Need for hospitalization or residence in a nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-07; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantine G. Lyketsos, MD, MHS, Study Chair — Johns Hopkins University
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina

REFERENCES:
- [Result] Rosenberg PB, Drye LT, Martin BK, Frangakis C, Mintzer JE, Weintraub D, Porsteinsson AP, Schneider LS, Rabins PV, Munro CA, Meinert CL, Lyketsos CG; DIADS-2 Research Group. Sertraline for the treatment of depression in Alzheimer disease. Am J Geriatr Psychiatry. 2010 Feb;18(2):136-45. doi: 10.1097/JGP.0b013e3181c796eb. PMID 20087081
- [Derived] Drye LT, Martin BK, Frangakis CE, Meinert CL, Mintzer JE, Munro CA, Porsteinsson AP, Rabins PV, Rosenberg PB, Schneider LS, Weintraub D, Lyketsos CG; DIADS-2 Research Group. Do treatment effects vary among differing baseline depression criteria in depression in Alzheimer's disease study +/- 2 (DIADS-2)? Int J Geriatr Psychiatry. 2011 Jun;26(6):573-83. doi: 10.1002/gps.2565. PMID 20672243
- [Derived] Martin BK, Frangakis CE, Rosenberg PB, Mintzer JE, Katz IR, Porsteinsson AP, Schneider LS, Rabins PV, Munro CA, Meinert CL, Niederehe G, Lyketsos CG. Design of Depression in Alzheimer's Disease Study-2. Am J Geriatr Psychiatry. 2006 Nov;14(11):920-30. doi: 10.1097/01.JGP.0000240977.71305.ee. PMID 17068314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from memory clinics at five academic centers in the United States.
Groups:
- Placebo: Participants will receive placebo matched to sertraline
  Placebo: Placebo designed to mimic sertraline taken daily for 24 weeks
- Sertraline: Participants will receive sertraline at a target dose of 100mg daily.
  Sertraline (Zoloft): Sertraline: range of 25 to 125 mg per day for 24 weeks
Period: Overall Study
Arm/Group | Placebo | Sertraline
Started | 64 | 67
Completed | 60 | 64
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 76.5 (8) | 78.2 (8) | 77.3 (8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 40 | 31 | 71
  Male | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Modfied Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (mADCS-CGIC)
Description: At each study visit, based on patient examination and caregiver interview, clinicians rated overall impression of clinical change from baseline using the modified Alzheimer's Disease Cooperative Study Clinical Global Impression of Change index (mADCS-CGIC), which in addition to the original scale incorporates a global rating of mood and associated symptoms of depression. The mADCS-CGIC uses a seven-point Likert scale, with scores ranging from 1 ("much better") to 7 ("much worse"), with a score of 4 being "no change".
Time Frame: Measured at Week 12
Measure: Number; unit: participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 67 | 64
participants
  "much worse" | 1 | 0
  "worse" | 5 | 2
  "a bit worse" | 6 | 9
  "no change" | 10 | 11
  "a bit better" | 18 | 18
  "better" | 18 | 21
  "much better" | 9 | 3
Statistical Analysis 1: Comparison: Sertraline vs Placebo; The statistical analyses compared data collected from the CGIC of participants who received sertraline who had a score equal to or better than the CGIC of participants who received the placebo intervention; Test type: Superiority or Other; p = 0.98, Chi-squared; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.52 to 1.97]

2. Secondary Outcome: Remission According to Cornell Scale for Depression in Dementia Scale
Description: The Cornell Scale for Depression in Dementia (CSDD), a 19-item scale measuring the severity of depression in dementia, utilizing input from both the caregiver and the participant. CSDD scores were imputed for 2 participants for week 2, 4 participants for week 4, 7 participants for week 8, and 12 participants for week 12.
Time Frame: Measured at Weeks 12
Measure: Number; unit: percentage of participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 67 | 64
percentage of participants | 33 | 19
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p = 0.11, Chi-squared; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.84 to 5.04]

ADVERSE EVENTS:
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 13/67 | 7/64
Other Adverse Events (participants affected / at risk) | 44/67 | 26/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=67) | Placebo (N=64)
Pneumonia/respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Neurologic (Nervous system disorders) | 4 | 3
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 | 1
Cardiac (Cardiac disorders) | 3 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=67) | Placebo (N=64)
Diarrhea (Gastrointestinal disorders) | 36 | 22
Dizziness (Nervous system disorders) | 44 | 26
Dry mouth (Respiratory, thoracic and mediastinal disorders) | 37 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No